CLINICAL TRIAL: NCT02651727
Title: A Phase 1 Study of VS-4718, a Focal Adhesion Kinase Inhibitor, in Combination With Nab-paclitaxel and Gemcitabine in Subjects With Advanced Cancer
Brief Title: Ph 1 Study of VS-4718, a FAK Inhibitor, in Combination With Nab-paclitaxel and Gemcitabine in Advanced Cancer Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the company's decision to de-prioritize 4718 development
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS-4718-103
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part B, Cohort 1- VS-4718, nab-paclitaxel, gemcitabine (Experimental): Part B, Cohort 1- IV treatment in 28-day cycles (nab-paclitaxel 125 mg/m2 over 30 minutes on Days 1, 8, and 15 and gemcitabine at 1000 mg/m2 over 30 minutes on Days 1, 8, and 15) and oral VS 4718 BID continuously starting on Day 1 of Cycle 1
  Interventions: Drug: Part B, Cohort 1- VS-4718, nab-paclitaxel, gemcitabine
- Part B, Cohort 2- VS-4718, nab-paclitaxel, gemcitabine (Experimental): Part B, Cohort 2- IV treatment for the first 2 cycles (nab-paclitaxel 125 mg/m2 over 30 minutes on Days 1, 8, and 15 and gemcitabine at 1000 mg/m2 over 30 minutes on Days 1, 8, and 15), followed by IV treatment and oral VS-4718 BID continuously starting on Day 1 of Cycle 3
  Interventions: Drug: Part B, Cohort 2- VS4718, nab-paclitaxel, gemcitabine
- Part A- VS-4718, nab-paclitaxel, gemcitabine (Experimental): Part A- intravenous (IV) treatment in 28-day cycles (nab-paclitaxel 125 mg/m2 over 30 minutes on Days 1, 8, and 15 and gemcitabine at 1000 mg/m2 over 30 minutes on Days 1, 8, and 15) and oral VS 4718 twice-daily (BID) continuously starting on Cycle 1 Day 2. The starting dose of VS-4718 will be 200 mg BID.
  Interventions: Drug: Part A- VS-4718, nab-paclitaxel, gemcitabine

INTERVENTIONS:
Drug: Part B, Cohort 1- VS-4718, nab-paclitaxel, gemcitabine — IV treatment in 28-day cycles (nab-paclitaxel 125 mg/m2 over 30 minutes on Days 1, 8, and 15 and gemcitabine at 1000 mg/m2 over 30 minutes on Days 1, 8, and 15) and oral VS 4718 BID continuously starting on Day 1 of Cycle 1
  Arms: Part B, Cohort 1- VS-4718, nab-paclitaxel, gemcitabine
Drug: Part B, Cohort 2- VS4718, nab-paclitaxel, gemcitabine — IV treatment for the first 2 cycles, followed by IV treatment and oral VS-4718 BID continuously starting on Day 1 of Cycle 3
  Arms: Part B, Cohort 2- VS-4718, nab-paclitaxel, gemcitabine
Drug: Part A- VS-4718, nab-paclitaxel, gemcitabine — Part A- intravenous (IV) treatment in 28-day cycles (nab-paclitaxel 125 mg/m2 over 30 minutes on Days 1, 8, and 15 and gemcitabine at 1000 mg/m2 over 30 minutes on Days 1, 8, and 15) and oral VS 4718 twice-daily (BID) continuously starting on Cycle 1 Day 2. The starting dose of VS-4718 will be 200 mg BID.
  Arms: Part A- VS-4718, nab-paclitaxel, gemcitabine

SUMMARY:
The purpose of this study is to evaluate increasing dose levels of VS-4718 administered in combination with gemcitabine and nab-paclitaxel in subjects with advanced cancer and to determine a recommended Phase 2 dose (RP2D) for further development of this combination in subjects with untreated advanced pancreatic cancer.

DETAILED DESCRIPTION:
The study is comprised of 2 sequential parts: Part A (Dose Escalation of VS-4718) in subjects with advanced cancer and Part B (Expansion) in subjects with untreated advanced pancreatic cancer.

Up to 60 evaluable subjects (i.e., subjects who complete at least 1 cycle (28 days) of therapy) will be enrolled, assuming that:

1. Part A: The maximum sample size will be 6 subjects up to 4 dose levels (exclusive of replacement subjects). However, additional subjects may be added if exploration of intermediate dose level(s) of VS 4718 is warranted. The starting dose of VS-4718 will be 200mg BID.
2. Part B: Up to 36 additional subjects may be enrolled at the RP2D. These subjects will be randomized at a 1:1 ratio to 1 of 2 treatment cohorts:

   * Cohort 1: IV treatment in 28-day cycles (nab-paclitaxel 125 mg/m2 over 30 minutes on Days 1, 8, and 15 and gemcitabine at 1000 mg/m2 over 30 minutes on Days 1, 8, and 15) and oral VS 4718 BID continuously starting on Day 1 of Cycle 1
   * Cohort 2: IV treatment for the first 2 cycles, followed by IV treatment and oral VS-4718 BID continuously starting on Day 1 of Cycle 3

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed diagnosis of an advanced nonhematological malignancy (Part A) or advanced pancreatic adenocarcinoma (Part B) that is not surgically resectable
* Eligible for treatment with nab-paclitaxel and gemcitabine on Days 1, 8, and 15 in 28-day cycles as standard therapy
* Evaluable or measurable disease, as assessed by RECIST v1.1
* ECOG performance status of ≤ 1
* Adequate renal function (creatinine ≤ 1.5×ULN [upper limit of normal]) or glomerular filtration rate of ≥ 60 mL/min
* Adequate hepatic function (total bilirubin ≤ 1.5×ULN for the institution; aspartate transaminase and alanine transaminase ≤ 2.5×ULN, or ≤ 5×ULN if due to liver involvement by tumor; albumin ≥ 3 g/dL)
* Adequate bone marrow function (hemoglobin ≥ 9.0 g/dL; unsupported platelets ≥ 100×109 cells/L; absolute neutrophil count [ANC] ≥ 1.5×109 cells/L without the use of hematopoietic growth factors)
* Corrected QT interval (QTc) < 470 ms
* Willing and able to participate in the trial and comply with all trial requirements

Exclusion Criteria:

* Gastrointestinal (GI) condition that could interfere with the swallowing or absorption of study medication
* Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases).
* History of upper gastrointestinal bleeding, ulceration, or perforation within 6 months prior to the first dose of protocol therapy
* Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of protocol therapy.
* Part B only: Prior therapy (including investigational agents) for pancreatic cancer
* Chemotherapy or radiotherapy within 14 days prior to first dose of protocol therapy
* Active treatment for a secondary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | 6 months
  Dose Escalation Phase: Frequency of DLTs at each dose level associated with administration of VS-4718 in combination with gemcitabine and nab-paclitaxel

SECONDARY OUTCOMES:
Progression Free Survival | From the date of first treatment to the date of progression including death from any cause, expected average at least 5 months
Response rate (RR) | Every 8 weeks from baseline through the end of treatment, an expected average of 5 months]
  RR is measured as the best overall response using Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1.
Pharmacokinetics of VS-4718 in combination with nab-paclitaxel and gemcitabine: Clearance | Time points on Day 1, 2,15, 16, and 22 in Cycle 1; Day 1 of each subsequent cycle
Pharmacokinetics of VS-4718 in combination with nab-paclitaxel and gemcitabine: Plasma concentration | Time points on Day 1, 2,15, 16, and 22 in Cycle 1; Day 1 of each subsequent cycle
Pharmacokinetics of VS-4718 in combination with nab-paclitaxel and gemcitabine: Area under the plasma concentration versus time curve (AUC) | Time points on Day 1, 2,15, 16, and 22 in Cycle 1; Day 1 of each subsequent cycle
Pharmacokinetics of VS-4718 in combination with nab-paclitaxel and gemcitabine: Maximum observed plasma concentration (Cmax) | Time points on Day 1, 2,15, 16, and 22 in Cycle 1; Day 1 of each subsequent cycle
Pharmacokinetics of VS-4718 in combination with nab-paclitaxel and gemcitabine: Time to reach maximum observed concentration (Tmax) | Time points on Day 1, 2,15, 16, and 22 in Cycle 1; Day 1 of each subsequent cycle
Pharmacokinetics of VS-4718 in combination with nab-paclitaxel and gemcitabine: Half life (T1/2) | Time points on Day 1, 2,15, 16, and 22 in Cycle 1; Day 1 of each subsequent cycle

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No